CLINICAL TRIAL: NCT06468644
Title: Phase II Study of Different Doses of Radiotherapy Combined With Sintilimab in the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ConES-ljc
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): dose 1 of radiotherapy+sintilimab
  Interventions: Drug: chemoradiotherapy （CRT）+sintilimab 1
- Group B (Experimental): dose 2 of radiotherapy+sintilimab
  Interventions: Drug: CRT+sintilimab 2

INTERVENTIONS:
Drug: chemoradiotherapy （CRT）+sintilimab 1 — radiotherapy (50.4Gy/1.8Gy/28f)+chemotherapy (paclitaxel 150mg/m2 D1+cisplatin 25mg/m2 D1-3，Q3W)+Sintilimab (200mg, iv, D1, Q3W) Consolidation therapy: Sintilimab: 200mg, iv, D1, Q3W
  Arms: Group A
Drug: CRT+sintilimab 2 — radiotherapy (60Gy/2Gy/30f)+chemotherapy (paclitaxel 150mg/m2 D1+cisplatin 25mg/m2 D1-3，Q3W)+Sintilimab (200mg, iv, D1, Q3W) Consolidation therapy: Sintilimab: 200mg, iv, D1, Q3W
  Arms: Group B

SUMMARY:
This study is aimed to evaluate the efficacy and safety of different doses of radiotherapy combined with sintilimab in locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study was designed as a two cohorts, phase II trial. Subjects will receive different doses of radiotherapy combined with sintilimab. The primary endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Histopathological examination of the primary biopsy confirmed the diagnosis of locally advanced esophageal squamous cell carcinoma
* At least one measurable lesion
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1
* With adequate organs function

Exclusion Criteria:

* Patients with active malignancy within 5 years other than the tumor studied in this study or a localized tumor that has been cured such as resected basal or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or breast cancer
* Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula
* Patients who have received any anti-tumor therapy for the research disease in the past, including radiotherapy, chemotherapy, immunotherapy (including but not limited to interleukin, interferon, thymus hormone) and traditional Chinese medicine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1 years
  the time from random assignment in a clinical trial to disease progression or death from any cause
Incidence rate of adverse events | 3 years
  The ratio of the number of cases with adverse events to the total number of cases available for evaluation.

SECONDARY OUTCOMES:
overall survival | 3 years
  the time from randomization to death
Objective Response Rate | 3 months after therapy
  the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors 1.1

IPD SHARING:
Plan to Share IPD: No